CLINICAL TRIAL: NCT07376135
Title: Digitally Supported Lifestyle Programme to Promote Brain Health Among Older Adults - the LETHE-AT Randomised-controlled, Multicentre Pilot Trial
Brief Title: LETHE-AT: a Personalized Multidomain Lifestyle Intervention for Individuals at Increased Risk of Memory Impairment.
Acronym: LETHE-AT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other); FH Joanneum Gesellschaft mbH (Industry); Medical University Innsbruck (Other); Austrian Research Promotion Agency (Other Government)
Responsible Party: Principal Investigator, Elisabeth Stögmann, Physician Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MUW EK Nr: 1792/2025; 58285128 / 921935 (Other Grant/Funding Number: Austrian Research Promotion Agency (FFG))
Record Dates: First submitted 2025-12-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD)
Keywords: dementia prevention; brain health; multidomain lifestyle intervention; Austria; multicenter; subjective cognitive decline; physical activity; cognitive training; wearable; smartwatch; App; risk reduction; randomized controlled trial; hybrid digital; dietary counselling; sleep; stress management; ANU-ADRI; LIBRA2; Neuropsychological Test Battery (NTB); telemedicine; Alzheimer Disease; Cognition Disorders; mild cognitive impairment; multimodal intervention; multicomponent intervention; motivational interviewing; health coaching; mHealth; eHealth
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Alzheimer Disease; Risk Reduction Behavior; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be actively told to what group they have been assigned (intervention or control). Outcome assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A self-guided multimodal lifestyle advice group (Sham Comparator): Participants in the control arm receive a self-guided lifestyle advice programme via the LETHE-AT app and smartwatch, with standardized information across all lifestyle domains but without motivational interviewing, structured coaching or algorithm-based personalization.
  Interventions: Behavioral: Self-guided multimodal lifestyle advice group
- A tailored hybrid multidomain lifestyle intervention group (Active Comparator): Participants in the intervention arm receive an MI-guided hybrid multidomain lifestyle intervention that integrates AI-based risk profiling, personalized goal setting and structured telehealth coaching with app- and smartwatch-supported self-management across six lifestyle domains.
  Interventions: Behavioral: A tailored hybrid multidomain lifestyle intervention group

INTERVENTIONS:
Behavioral: A tailored hybrid multidomain lifestyle intervention group — The structured counselling intervention combines interactive face-to-face workshops with ongoing remote coaching through the LETHE-AT mobile app and regular (video)-telephone sessions to support sustained lifestyle changes. Each participant is individually guided throughout the intervention by a dedicated coach (physician or psychologist), trained in motivational interviewing techniques aimed at facilitating behavioural changes across targeted lifestyle domains.
  Arms: A tailored hybrid multidomain lifestyle intervention group
Behavioral: Self-guided multimodal lifestyle advice group — Participants receive a reduced version of the LETHE-AT app with general health information only. No structured in-person or remote counselling is provided and no individualized digital content is unlocked. They are encouraged to implement lifestyle changes independently. Throughout the trial, participants complete the same in-app questionnaires, wear a Garmin Vivosmart 5, and receive routine laboratory result with advice to seek certain medical care if needed. A pure no-treatment arm is not included for ethical reasons.
  Arms: A self-guided multimodal lifestyle advice group

SUMMARY:
The goal of this clinical trial is to learn whether a hybrid multidomain lifestyle program can prevent cognitive decline and reduce dementia risk in community-dwelling adults in mid- to late life who are at increased risk of Alzheimer´s disease or related dementias but do not yet have significant cognitive impairment.

The main question the study aims to answer are:

* Whether the structured hybrid multidomain lifestyle intervention is feasible (e.g., adherence and retention rate), and how well the digital components are accepted and implemented in the intervention group.
* Does the intervention reduces the overall burden of modifiable dementia risk factors and improves global cognitive performance compared with usual care.

Researchers will compare participants assigned to the tailored hybrid multidomain lifestyle intervention group with those in a self-guided multimodal lifestyle advice group.

Participants assigned to the intervention group will receive a plan adjusted to their individual dementia risk profile. A physician trained in motivational interviewing will review their progress continuously.

The self-guided multimodal lifestyle advice group will receive rigid but comprehensible lifestyle health advice with reduced access to digital support tools.

Participants will:

* Complete an initial risk assessment that uses machine-learning triage to identify and prioritize their most important modifiable dementia risk factors.
* Receive personalized recommendations for gradual lifestyle change, including physical activity, nutrition, cognitive training, other dementia risk-factor management (e.g. hearing impairment), stress & sleep management, and social activities.
* Use a smartphone and smartwatch to passively collect digital biomarkers and to complete questionnaires at regular intervals, so that physicians trained in motivational interviewing can adapt goals through shared decision making.
* Use a study app as the central access point for the program, including educational content, progress tracking, and gamified challenges with social comparison and incentives.

DETAILED DESCRIPTION:
LETHE AT is an 18 month multicentre randomized controlled trial in Austria that evaluates a tailored hybrid multidomain lifestyle intervention programme in older adults with multiple dementia risk factors and is conducted at the Medical Universities of Vienna, Innsbruck, and Graz.

Previous multidomain lifestyle trials have shown that structured interventions targeting modifiable risk factors can attenuate cognitive decline and reduce dementia risk. These programme have used different delivery formats, including intensive face to face interventions (FINGER), fully digital approaches (Maintain Your Brain), and hybrid models (SMART and LETHE EU). LETHE-AT builds on this foundation by combining refined risk profiling and motivational interviewing (MI) with a centrally organized online and telephone prescreening process. This approach identifies cognitively unimpaired adults with a high burden of dementia risk factors and reduces avoidable on-site screening failures and participant disappointment.

Following the prescreening, comprehensive on-site screening is conducted at three Austrian memory clinics to enroll 300 participants. Eligibility is determined using predefined inclusion and exclusion criteria, including age 55-75 years, preserved cognition, subjective cognitive decline or a first-degree family history of dementia, the presence of at least three of 14 established modifiable dementia risk factors (e.g. hearing impairment, elevated LDL cholesterol), and sufficient motivation for lifestyle change as evaluated by physicians trained in MI.

Eligible participants are invited for a baseline visit, where dementia risk is quantified using LIBRA2 and ANU-ADRI, and a harmonized neuropsychological and functional assessment battery is administered by trained neuropsychologists.

The study population is then stratified by sex, age and study site and randomly assigned in a 1:1 ratio to the tailored hybrid multidomain lifestyle intervention group or to the self-guided multimodal lifestyle advice group.

At a subsequent in-person visit, all participants attend a structured onboarding session. In both groups, the smartphone, smartwatch and LETHE-App are introduced, standardized usage instructions are provided, and access to ongoing technical support is ensured.

In the MI-guided hybrid multidomain lifestyle intervention group, onboarding additionally includes an individual consultation with a trained MI-coach.

The 14 modifiable risk factors are mapped onto six lifestyle domains (diet, physical activity, cognitive engagement, sleep and stress, social interactions, and other risk-factor management) to guide content and provide a replicable coaching framework. Additionally, the modifiable risk profile is processed by a dedicated AI-based decision-support tool that generates tailored goal recommendations, and a complemental questionnaire captures personal preferences and constraints. Based on this information, participants and the MI coach select personal goals from a predefined list, with each goal allocated to one of the six lifestyle domains.

The intervention programme begins with a small set of high-priority goals and is gradually expanded, with the number and intensity of goals adapted over time to each participant's risk profile, capacity and circumstances. The intervention programme is harmonized across study sites and supported by manuals to ensure consistent delivery.

The LETHE-App is provided to both study arms and serves several purposes. First, it enables continuous assessment of digital markers (e.g., log-in patterns), complemented by digital biomarkers from the smartwatch (e.g., sleeping-time). Second, it delivers frequent questionnaires on system satisfaction and risk-factor status. In addition, the app offers reminders and review functions for personal goals and provides evidence-based lifestyle information for each domain, including content supplied by the Austrian Agency for Health and Food Safety (AGES). Further functions, such as gamification elements to support adherence and motivation to change, are planned for iterative development.

Participants attend in-person study visits at baseline, month 9 and month 18, where they undergo an extended neuropsychological test battery, standardized dementia risk assessment and blood sampling. Brain MRI is performed as part of an imaging sub-study, and blood samples are stored for analysis of conventional risk markers and exploratory dementia-related biomarkers.

Outcome assessors for cognition, imaging and laboratory measures are blinded to group allocation, and group assignment is not revealed in study documentation used for these assessments.

Intervention study visits consist of individual MI-based tele-health sessions of approximately 20 to 30 minutes, scheduled at roughly three-month intervals to review progress, troubleshoot barriers and adjust goals. A harmonized protocol is used across sites, and sessions focus on strengthening intrinsic motivation for lifestyle change by exploring ambivalence, linking behaviour change to personally meaningful values and reinforcing self-efficacy in initiating and maintaining lifestyle modifications.

Safety is monitored through brief adverse event questionnaires at scheduled time points and through spontaneous reports during visits or phone contacts. All study related events are documented and managed according to protocol, and the intervention is nonpharmacologic and consistent with current dementia prevention guidelines. Data are pseudonymized and stored on secure servers with restricted access and audit trails, and trial conduct follows Good Clinical Practice and standardized operating procedures with trained staff and a central data management plan.

The planned sample of 300 participants reflects the focus on feasibility outcomes such as counseling acceptability, adherence and retention. Analyses follow the intention to treat principle and use linear mixed effects models with group, time and their interaction adjusted for baseline values and prespecified covariates. Effect estimates are reported with 95 percent confidence intervals, and missing data are examined in planned sensitivity analyses. No formal interim efficacy analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 75 years at the time of screening.
* Fluency in German.
* All participants must be able and willing to provide written informed consent form (ICF) prior to any study-related procedures.
* Ownership of a compatible Android smartphone, or willingness and capability to use a study-provided Android smartphone for the duration of the study.
* Subjective cognitive decline and/or a positive first-degree family history of dementia.
* Willingness to make meaningful changes in at least three of six lifestyle domains: dietary counselling, physical activity, cognitive training, vascular risk management, social interaction, and sleep and relaxation.
* Cognitive performance at or slightly below age expectations, defined as an m-TICS (modified Telephone Interview for Cognitive Status) score ≥ 37/50, and a Montreal Cognitive Assessment (MoCA) ≥ 26/30.

Exclusion Criteria:

* Diagnosed or suspected dementia or substantial cognitive impairment, defined as an m-TICS score ≤ 36 or MoCA < 26, or current or previous use of Alzheimer´s disease or other dementia medication.
* Significant neurological disease, including but not limited to Parkinson´s disease, Huntington´s disease, normal pressure hydrocephalus, brain tumour, progressive supranuclear palsy, seizure disorder, subdural haematoma, multiple sclerosis, or a history of significant head trauma with persistent neurological sequelae or known structural brain abnormalities.
* Diminished decision-making capacity, inability to provide informed consent, inability to complete study assessments, or any condition preventing effective cooperation, as determined by clinical judgement.
* Severe impairment of vision, hearing, or communication abilities that would preclude participation in study procedure.
* Any medical or psychiatric condition affecting safe engagement, including but not limited to active malignancy, major depressive disorder, symptomatic cardiovascular disease, or revascularisation procedures within the past year.
* Current participation in another interventional trial, unless the study team determines this does not interfere with participation in the LETHE-AT.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Operational feasibility: retention rate | Baseline to 18 months
  Proportion of all randomized participants who complete the Month 18 assessment in each trial arm (percentage of all randomized participants; higher percentage = better retention).
Operational feasibility: adherence to the structured hybrid lifestyle intervention | Continuously assessed over 18 months
  Composite adherence score combining attendance at workshops and telehealth sessions, engagement with the LETHE-AT app (logins and completed modules), and proportion of days with successful smartwatch data uploads (higher values = better adherence).

SECONDARY OUTCOMES:
Change in health-related quality of life (SF-36) | Baseline to 18 months
  Change in health-related quality of life assessed with the 36-Item Short Form Health Survey (SF-36; 0-100 points per domain; higher scores = better self-reported health status).
Change in health literacy (HLS-EU-Q16) | Baseline to 18 months
  Change in health literacy assessed with the European Health Literacy Survey Questionnaire, 16-item version (HLS-EU-Q16; 0-16 points; higher scores = better general health literacy).
User acceptance of the digital solution (SUS) | 2 months past enrollment to 18 months
  Change in perceived usability of the app and digital devices assessed with the System Usability Scale (SUS; 0-100 points; higher scores = better perceived usability and acceptance).
Change in perceived stress (PSS-14) | Baseline, Month 9, 18 months.
  Change in perceived stress assessed with the Perceived Stress Scale-14 (PSS-14; 0-56 points; higher scores = more perceived stress during the past month).
Change in insomnia symptoms (ISI) | Baseline, Month 9, 18 months
  Change in insomnia symptoms assessed with the Insomnia Severity Index (ISI; 0-28 points; higher scores = more severe insomnia complaints).

OTHER OUTCOMES:
Change in global cognition assessed with the modified Neuropsychological Test Battery (mNTB) | Baseline (Month 0) to Month 18.
  All test raw scores are converted to z-scores (baseline mean = 0, SD = 1, with sign reversal where lower times indicate better performance):
  Wechsler Memory Scale - Fourth Edition (WMS-IV) Logical Memory (immediate and delayed recall, recognition)
  Rey Auditory Verbal Learning Test (RAVLT / VLMT; list learning, immediate and delayed recall, recognition)
  Rey-Osterrieth Complex Figure Test (copy, 3-minute and 30-minute delayed recall)
  Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span (forward, backward, sequencing)
  Test of Attentional Performance (TAP) - Alertness
  Test of Attentional Performance (TAP) - Divided Attention
  WAIS-IV Digit Symbol Substitution Test (DSST)
  Trail Making Test (TMT) Part A
  Trail Making Test (TMT) Part B (shitime B-A)
  Regensburg Word Fluency Test (semantic: animals; phonemic: letter P)
  Colour-Word Interference Test (German Stroop; colour naming, word reading, interference condition)
Change in dementia risk: LIBRA2 | Baseline and Month 18.
  Change in dementia risk estimated with the Lifestyle for Brain Health index (LIBRA2; theoretical range -5.9 to +12.7; higher scores = less healthy lifestyle and higher estimated dementia risk).
Change in dementia risk: ANU-ADRI | Baseline and Month 18.
  Change in dementia risk estimated with the Australian National University Alzheimer's Disease Risk Index (ANU-ADRI; theoretical range approximately -13 to +64; higher scores = higher estimated Alzheimer's disease risk).
Change in physical activity (German-PAQ) | Baseline, Month 9, Month 18.
  Change in self-reported physical activity assessed with the Short German Physical Activity Questionnaire (German-PAQ; minutes per week of moderate-to-vigorous activity; higher values = more physical activity).
Change in depressive symptoms (SDS) | Baseline, Month 9, Month 18
  Change in depressive symptoms assessed with the Zung Self-Rating Depression Scale (SDS; 20-80 points; higher scores = more depressive symptom burden).
Change in Mediterranean diet adherence (MEDAS) | Baseline, Month 9, Month 18
  Change in diet quality assessed with the 14-Item Mediterranean Diet Adherence Screener (MEDAS; 0-14 points; higher scores = better adherence to a Mediterranean-style diet).
Change in functional abilities (FAQ) | Baseline, Month 9, Month 18
  Change in instrumental activities of daily living assessed with the Functional Activities Questionnaire (FAQ; 0-30 points; higher scores = greater functional impairment in IADL).
Change in social engagement (LSNS-6) | Baseline, Month 9, Month 18
  Change in social networks assessed with the Lubben Social Network Scale-6 (LSNS-6; 0-30 points; higher scores = larger and more supportive social network).
Change in cognitive reserve (CRQi) | Baseline, Month 9, Month 18
  Change in cognitive reserve assessed with the Cognitive Reserve questionnaire index. (higher scores = greater lifetime cognitive reserve from education and stimulating activities)
Change in physical functioning (SPPB and grip strength) | Baseline, Month 9, Month 18
  Change in lower-extremity function assessed with the Short Physical Performance Battery (SPPB; 0-12 points; higher scores = better balance, gait and chair-rise performance) and change in hand grip strength measured in kilograms with a dynamometer.
Change in smoking dependence (FTND) | Baseline, Month 9, Month 18
  Change in nicotine dependence among current smokers assessed with the Fagerström Test for Nicotine Dependence (FTND; 0-10 points; higher scores = stronger nicotine dependence).
Change in alcohol consumption (AUDIT-C) | Baseline, Month 9, Month 18
  Change in alcohol use assessed with the Alcohol Use Disorders Identification Test - Consumption subscale (AUDIT-C; 0-12 points; higher scores = higher risk of hazardous drinking).
Change in AD-related blood biomarkers | Baseline and Month 18 (subsample).
  Change in plasma Aβ42/40 ratio, phosphorylated tau (e.g. p-tau217) and neurofilament light chain (NfL) as markers of Alzheimer-related and neuroaxonal pathology (higher levels = greater pathology).
Ten-year cardiovascular disease risk (Framingham Risk Score) | Baseline and Month 18.
  Change in 10-year cardiovascular risk estimated using the Framingham Risk Score (percentage probability based on age, blood pressure, lipids, smoking and diabetes status; higher values = higher predicted CVD risk).
Change in attitudes towards dementia risk reduction (selected MCLHB-DRR items) | Baseline, 9 Months, 18 Months
  Change in participants' motivation, perceived benefits, and perceived personal relevance of dementia risk reduction, assessed with selected items from the MCLHB-DRR scale (higher scores indicating more positive attitudes towards adopting risk-reducing behaviours).
Change in hippocampal volume (MRI) | Near Baseline and near Month 18 (±2 months; optional MRI sub study)
  Change in hippocampal volume measured on high resolution structural MRI.
Change in cortical thickness (MRI) | Near Baseline and near Month 18 (±2 months; optional MRI sub study)
  Change in cortical thickness measured on high resolution structural MRI.
Change in white matter integrity (MRI) | Near Baseline and near Month 18 (±2 months; optional MRI sub study)
  Change in white matter integrity measured on diffusion weighted MRI.
Change in resting state connectivity indices (MRI) | Near Baseline and near Month 18 (±2 months; optional MRI sub study)
  Change in resting state connectivity indices measured on resting state functional MRI.
Change in resting heart rate (Continuously) | Continuously for 18 months.
  Change in resting heart rate derived from continuous wrist photoplethysmography recorded day and night by the Garmin Vivosmart 5 smartwatch.
Change in Sleep Score (Continuously) | Continuously for 18 months.
  Change in Sleep Score derived from wearable identified sleep stages combined into a single Sleep Score (Garmin Vivosmart 5).
Change in minutes of moderate to vigorous activity (Continuously) | Continuously for 18 months.
  Change in minutes of moderate to vigorous activity captured by the Garmin Vivosmart 5 smartwatch.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medical University of Innsbruck, Graz, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including baseline characteristics, primary and key secondary outcomes) underlying the main published results will be made available to qualified researchers upon reasonable request, after approval by the sponsor and the relevant ethics committees.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be made available after publication of the primary results for a limited period to be specified in the final data sharing policy.
Access Criteria: Access will be granted to qualified researchers upon reasonable request and subject to sponsor and ethics committee approval, according to the final data sharing policy.
URL: https://www.lethe.at/

REFERENCES:
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Yaffe K, Vittinghoff E, Dublin S, Peltz CB, Fleckenstein LE, Rosenberg DE, Barnes DE, Balderson BH, Larson EB. Effect of Personalized Risk-Reduction Strategies on Cognition and Dementia Risk Profile Among Older Adults: The SMARRT Randomized Clinical Trial. JAMA Intern Med. 2024 Jan 1;184(1):54-62. doi: 10.1001/jamainternmed.2023.6279. PMID 38010725
- [Background] Brodaty H, Chau T, Heffernan M, Ginige JA, Andrews G, Millard M, Sachdev PS, Anstey KJ, Lautenschlager NT, McNeil JJ, Jorm L, Kochan NA, Maeder A, Welberry H, San Jose JC, Briggs NE, Popovic G, Mavros Y, Almendrales Rangel C, Noble Y, Radd-Vagenas S, Flood VM, O'Leary F, Lampit A, Walton CC, Barr P, Fiatarone Singh M, Valenzuela M. An online multidomain lifestyle intervention to prevent cognitive decline in at-risk older adults: a randomized controlled trial. Nat Med. 2025 Feb;31(2):565-573. doi: 10.1038/s41591-024-03351-6. Epub 2025 Jan 28. PMID 39875685
- [Background] Frisoni GB, Altomare D, Ribaldi F, Villain N, Brayne C, Mukadam N, Abramowicz M, Barkhof F, Berthier M, Bieler-Aeschlimann M, Blennow K, Brioschi Guevara A, Carrera E, Chetelat G, Csajka C, Demonet JF, Dodich A, Garibotto V, Georges J, Hurst S, Jessen F, Kivipelto M, Llewellyn DJ, McWhirter L, Milne R, Minguillon C, Miniussi C, Molinuevo JL, Nilsson PM, Noyce A, Ranson JM, Grau-Rivera O, Schott JM, Solomon A, Stephen R, van der Flier W, van Duijn C, Vellas B, Visser LNC, Cummings JL, Scheltens P, Ritchie C, Dubois B. Dementia prevention in memory clinics: recommendations from the European task force for brain health services. Lancet Reg Health Eur. 2023 Jan 31;26:100576. doi: 10.1016/j.lanepe.2022.100576. eCollection 2023 Mar. PMID 36895446
- [Background] Schulz CP, Claas P, Stienkemeier F. Formation of K*He exciplexes on the surface of helium nanodroplets studied in real time. Phys Rev Lett. 2001 Oct 8;87(15):153401. doi: 10.1103/PhysRevLett.87.153401. Epub 2001 Sep 21. PMID 11580696
- [Background] Livingston G, Huntley J, Liu KY, Costafreda SG, Selbaek G, Alladi S, Ames D, Banerjee S, Burns A, Brayne C, Fox NC, Ferri CP, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Nakasujja N, Rockwood K, Samus Q, Shirai K, Singh-Manoux A, Schneider LS, Walsh S, Yao Y, Sommerlad A, Mukadam N. Dementia prevention, intervention, and care: 2024 report of the Lancet standing Commission. Lancet. 2024 Aug 10;404(10452):572-628. doi: 10.1016/S0140-6736(24)01296-0. Epub 2024 Jul 31. No abstract available. PMID 39096926